CLINICAL TRIAL: NCT02140463
Title: Next Generation pErsonalized tX(Therapy) With Plasma DNA Trial-2 in Refractory Solid Tumors (The NEXT-2 Trial)
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, Professor, Samsung Medical Center
Other Study IDs: 2013-11-014
Record Dates: First submitted 2014-02-10; First posted 2014-05-16 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Metastatic Gastrointestinal Cancer; Genitourinary Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms; Urogenital Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — circulating free DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- metastatic cancer: metastatic gastrointestinal cancer metastatic genitourinary cancer other rare cancer lung cancer

SUMMARY:
Analysis of cell free DNA(cfDNA), unlike tissue biopsy, presents a new tool for the monitoring and treatment of cancer. The investigators have developed a differentiated sequencing assay, Digital Sequencing Technology (DST) that enables detection of rare genomic abnormalities with ultra high-specificity and sensitivity. The investigators assay is able to eliminate the error and distortion created by sample-prep and sequencing processes in standard NGS(next-generation sequencing ) workflows and produce near-perfect representations of all rare variants.

The investigators have shown that in sequencing a comprehensive cancer panel of 80kbp in 0.1% cancer cell line titration samples, standard Illumina SBS(sequencing by synthesis ) generates many high-quality false positive variant calls in the range of 0.05-5%, while the investigators assay resulted in highly sensitive and completely error-free variant calls across the entire panel.

This work indicates the remarkable potential of using the investigators assay in deep analysis of cfDNA, thereby allowing researchers and clinicians to comprehensively and non-invasively monitor the genetic dimension of cancer throughout the body.

DETAILED DESCRIPTION:
Same as above

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 20 years
* Patients with histologically confirmed metastatic gastrointestinal cancer, rare cancer, lung cancer
* Patients with histologically confirmed metastatic cancer, who do not have sufficient biopsy material to undergo mutational testing of their tumor, or do not have feasible biopsy sites; melanoma/lung cancer and any solid tumor cancer types will be eligible for the study.
* Written informed consent form

Exclusion Criteria:

* Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical condition that would interfere with the subject's safety.
* Double primary cancer (except for any cancer in remission for > 5 years, cervix cancer in situ, basal cell cancer in situ, any in situ cancers that are resected)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pathologically confirmed cancer patient
Sampling Method: Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
feasibility | From date of start of targeted treatment oriented by NEXT until the date of first progression or date of death from any cause, whichever came first, assessed up to 1 year ]
  The feasibility of the use of plasma cell free DNA - molecular profiling to direct targeted therapies in the treatment of refractory solid tumors
  -ANALYSIS : The analysis of this exploratory study will be primarily descriptive. Data will be presented by means of summary statistics tables, graphs and listings.

SECONDARY OUTCOMES:
progression free survival (PFS), | 1years
  The progression free survival (PFS), duration of response and overall survival of patients with refractory solid tumors.
molecular profile with cell-free DNA | From date of start of targeted treatment oriented by NEXT until the date of first progression or date of death from any cause, whichever came first, assessed up to 1 year ]
  To compare the correlation between primary/metastatic tumor formalin-fixed paraffin-embedded DNA molecular profile with cell-free DNA from plasma
serial cfDNA samples | From date of start of targeted treatment oriented by NEXT until the date of first progression or date of death from any cause, whichever came first, assessed up to 1 year ]
  To evaluate changes in the tumor's molecular profile on serial cfDNA samples when patients progress after an initial response to targeted treatment
Duration of response | 1years
  The progression free survival (PFS), duration of response and overall survival of patients with refractory solid tumors.
overall survival | 1years
  The progression free survival (PFS), duration of response and overall survival of patients with refractory solid tumors.
response rate | up to 1 year
  The response rate of molecular-profile directed treatments in refractory solid tumors

CONTACTS AND LOCATIONS:
Overall Officials: Won Ki Kang, MD, Study Chair — Division of Hematology-Oncology, Department of Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, Korea
Locations (1):
- Samsung Medical Center, Seoul, South Korea